CLINICAL TRIAL: NCT01043926
Title: A Single Dose Study to Investigate the Pharmacokinetics of MK-4305 in Patients With Hepatic Insufficiency
Brief Title: Pharmacokinetics of Suvorexant in Participants With Hepatic Insufficiency (MK-4305-017)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4305-017; 2010_500 (Other: Merck Registration Number)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Insomnia; Hepatic Insufficiency
Keywords: Hepatic Insufficiency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hepatic Insufficiency | interventions — suvorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Participants with Moderate Hepatic Insufficiency (Part I) (Experimental): Participants with moderate hepatic insufficiency will receive a single dose of 20 mg open-label suvorexant during Part I of the study.
  Interventions: Drug: Suvorexant
- Healthy Participants (Part I) (Experimental): Healthy participants matched to participants with moderate hepatic insufficiency will receive a single dose of 20 mg open-label suvorexant during Part I of the study.
  Interventions: Drug: Suvorexant
- Participants with Mild Hepatic Insufficiency (Part II) (Experimental): Participants with mild hepatic insufficiency will receive a single dose of 20 mg open-label suvorexant during Part II of the study (if conducted).
  Interventions: Drug: Suvorexant
- Healthy Participants (Part II) (Experimental): Healthy participants matched to participants with mild hepatic insufficiency will receive a single dose of 20 mg open-label suvorexant during Part II of the study (if conducted).
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — single 20 mg dose of suvorexant will be administered as 2 x 10 mg film coated tablets on Day 1 after an overnight fast with water.
  Other Names: MK-4305

SUMMARY:
This study will determine whether the plasma concentration-time profile and pharmacokinetics (PK) of suvorexant (MK-4305) in participants with moderate and mild hepatic insufficiency are similar to those observed in healthy participants.

DETAILED DESCRIPTION:
Study Design:

This study plans to enroll 16 participants in Part I (8 participants with moderate hepatic insufficiency and 8 healthy participants) and 16 participants in Part II (8 participants with mild hepatic insufficiency and 8 healthy participants).

Part II will be conducted only if the primary hypothesis is not met and there is a significant difference in the PK of suvorexant between healthy participants and moderate hepatic insufficiency participants in Part I.

ELIGIBILITY:
Inclusion Criteria for Hepatic Insufficiency Participants:

* Females of reproductive potential must have a negative pregnancy test and agree to use (and/or have their partner use) two acceptable methods of birth control
* Body Mass Index (BMI) ≤35 kg/m^2 prior to start of study
* Diagnosis of stable hepatic insufficiency
* Smoking is restricted to ≤10 cigarettes per day

Inclusion Criteria for Healthy Matched Participants:

* Females of reproductive potential must have a negative pregnancy test and agree to use (and/or have their partner use) two acceptable methods of birth control
* BMI within approximately 20% of that of his/her hepatic participant
* Participant is healthy
* Participant is matched by race, gender, age (+/- 5 yrs) to his/her hepatic participant enrolled in the study
* Smoking is restricted to ≤10 cigarettes per day

Exclusion Criteria for Hepatic Insufficiency Participants:

* Participant is mentally or legally incapacitated
* History of a clinically significant psychiatric disorder over the last 5 to 10 years
* Participant has a history of any illness not related to his/her hepatic insufficiency
* History of a persistent sleep abnormality occurring for at least three (3)

months

* Participant has a history of stroke, chronic seizures, or major neurological disorder
* History of clinically significant hematological, immunological, renal,

respiratory, or genitourinary abnormalities, uncomplicated kidney stones or childhood asthma

* History of cancer
* History of cataplexy
* Participant is a nursing mother
* Participant consumes >3 servings of alcohol a day
* Participant consumes >6 caffeine servings a day
* History of multiple and/or severe allergies
* Participant is currently using or has history of illegal drug use
* Participant has traveled across 3 or more time zones within 2 weeks of study participation
* Participant works a night shift and is not able to avoid night shift work within 1 week before each treatment visit

Exclusion Criteria for Healthy Matched Participants:

* Participant is mentally or legally incapacitated. History of a clinically significant psychiatric disorder over the last 5 to 10 years.
* Participant has a history of any illness
* History of a persistent sleep abnormality occurring for at least three (3) months
* Participant has a history of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal,

cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities, uncomplicated kidney stones or childhood asthma

* History of cancer
* History of cataplexy
* Participant is a nursing mother
* Participant consumes >3 servings of alcohol a day
* Participant consumes >6 caffeine servings a day
* History of multiple and/or severe allergies
* Participant is currently using or has history of illegal drug use
* Participant has a history of any chronic and/or active hepatic disease
* Participant has traveled across 3 or more time zones within 2 weeks of study participation
* Participant works a night shift and is not able to avoid night shift work within 1 week before each treatment visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02-22 (Actual); Primary Completion 2010-04-14 (Actual); Study Completion 2010-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-017&kw=4305-017&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were enrolled in Part I of the study. Because the primary hypothesis was met, no participants were enrolled in Part II of the study.
Groups:
- Participants With Moderate Hepatic Insufficiency (Part I): Participants with moderate hepatic insufficiency received a single dose of 20 mg open-label suvorexant.
- Healthy Participants (Part I): Healthy participants matched to participants with moderate hepatic insufficiency received a single dose of 20 mg open-label suvorexant.
- Participants With Mild Hepatic Insufficiency (Part II): Participants with mild hepatic insufficiency were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled on this arm.
- Healthy Participants (Part II): Healthy participants matched to participants with mild hepatic insufficiency were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled on this arm.
Period: Overall Study
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I) | Participants With Mild Hepatic Insufficiency (Part II) | Healthy Participants (Part II)
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only presented for participants in Part I of the study (N=16). No participants were enrolled in Part II of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (5.1) | 57 (4.0) | 57.3 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to Infinity (0-∞) After Single Dose Suvorexant: Moderate Hepatic Insufficiency Participants Versus Healthy Participants (Part I)
Description: Overall exposure was assessed by the area under the plasma concentration versus time curve from time zero to infinity (AUC[0-∞]). AUC(0-∞) was calculated as the sum of the AUC to the last time point with a detectable plasma concentration (AUC[0-last]) and Ct/λ, where Ct was the last measurable concentration and λ was the apparent terminal rate constant.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Population: All Treated Participants
Measure: Geometric Mean (95% Confidence Interval); unit: μM•hr
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
μM•hr | 14.09 [10.48 to 18.93] | 13.73 [10.09 to 18.69]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Insufficiency (Part I) vs Healthy Participants (Part I); The geometric mean (GM) for each participant group and the corresponding 95% confidence interval (CI) were calculated for AUC(0-∞) using an analysis of covariance (ANCOVA) model. The AUC(0-∞) geometric mean ratio (GMR) of the 2 participant groups was used to test the primary hypothesis, which was that the AUC(0-∞) of suvorexant following a single 20-mg oral dose would be similar between participants with moderate hepatic insufficiency and healthy matched control participants; Test type: Non-Inferiority or Equivalence — AUC(0-∞) GMR = AUC(0-∞) GM for Moderate Hepatic Insufficiency Participants ÷ AUC(0-∞) GM for Healthy Participants A 90% CI for the AUC(0-∞) GMR was computed from the ANCOVA model. As prespecified by the analysis plan, if the upper limit bound of the 90% CI for the AUC(0-∞) GMR fell below 2.00, then the hypothesis would be met and the AUC(0-∞) of suvorexant would be similar in both groups of participants. That is, if the true ratio of the GM AUC(0-∞) is no more than 2.00; ANCOVA; AUC(0-∞) Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.74 to 1.43]

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Suvorexant After Single Dose: Moderate Hepatic Insufficiency Participants Versus Healthy Participants
Description: Cmax was defined as the maximum observed concentration of a drug after administration.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Population: All Treated Participants
Measure: Geometric Mean (95% Confidence Interval); unit: μM
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
μM | 0.800 [0.603 to 1.062] | 0.854 [0.636 to 1.147]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Insufficiency (Part I) vs Healthy Participants (Part I); The GM for each participant group and the corresponding 95% CI were calculated for Cmax using an ANCOVA model. The Cmax GMR of the 2 participant groups was used to test the primary hypothesis, which was that the Cmax of suvorexant following a single 20-mg oral dose would be similar between participants with moderate hepatic insufficiency and healthy matched control participants; Test type: Non-Inferiority or Equivalence — Cmax GMR = Cmax GM for Moderate Hepatic Insufficiency Participants ÷ Cmax GM for Healthy Participants A 90% CI for the Cmax GMR was computed from the ANCOVA model. As prespecified by the analysis plan, if the upper limit bound of the 90% CI for the Cmax GMR fell below 2.00, then the hypothesis would be met and the Cmax of suvorexant would be similar in both groups of participants. That is, if the true ratio of the geometric mean Cmax is no more than 2.00; ANCOVA; Cmax Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.68 to 1.29]

3. Primary Outcome: AUC(0-∞) After Single Dose Suvorexant: Mild Hepatic Insufficiency Participants Versus Healthy Participants (Part II)
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Population: Per protocol, the decision to perform AUC(0-∞) analysis in mild hepatic insufficiency participants was conditional on results of AUC(0-∞) analysis in moderate hepatic insufficiency participants. Since the primary hypothesis in moderate hepatic insufficiency participants was met, AUC(0-∞) analysis in mild hepatic insufficiency was not done.
Groups:
- Participants With Mild Hepatic Insufficiency (Part II): Participants with mild hepatic insufficiency were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
- Healthy Participants (Part II): Healthy participants matched to participants with mild hepatic insufficiency were to receive a single dose of 20 mg open-label suvorexant during Part II of the study. No participants were enrolled in this arm.
Arm/Group | Participants With Mild Hepatic Insufficiency (Part II) | Healthy Participants (Part II)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug.
Time Frame: From administration of study drug through 14 days after administration of study drug
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
participants | 7 | 5

5. Secondary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 4
Time Frame: From administration of study drug through 14 days after administration of study drug
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I)
Number analyzed (Participants) | 8 | 8
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study drug administration up to approximately 14 days post study drug administration.
Arm/Group | Participants With Moderate Hepatic Insufficiency (Part I) | Healthy Participants (Part I)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Moderate Hepatic Insufficiency (Part I) (N=8) | Healthy Participants (Part I) (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Somnolence (Nervous system disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.